CLINICAL TRIAL: NCT03476031
Title: Different Histopathological Patterns in Patients With HCV Nephropathy
Brief Title: Pathology of Hepatitis c Nephropathy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mahmoud Essmat Mohammad, principal investigator, Assiut University
Other Study IDs: DHPP
Record Dates: First submitted 2018-03-18; First posted 2018-03-23 (Actual); Last update posted 2018-03-23 (Actual); Status verified 2018-03

CONDITIONS: Cryoglobulinaemia Due to Chronic Hepatitis C

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- study group: patients with hepatitis c nephropathy detected by lab and renal biopsy
  Interventions: Diagnostic Test: renal biopsy

INTERVENTIONS:
Diagnostic Test: renal biopsy — needle biopsy will be taken from the kidney tissue then, diagnosed

SUMMARY:
Hepatitis c associated glomerulonephritis is an immune complex disease that occurs in 21% of patients who have HCV infection.

DETAILED DESCRIPTION:
Hepatitis C virus infection is a major public health problem with an estimated global prevalence of 3% and an estimated 5-20% of infected patients will develop liver cirrhosis .The Prevalence of Hepatitis C infection in end stage renal disease is greater than in the general population especially in those on hemodialysis which reflects nosocomial transmission of the disease in the hemodialysis environment.

Hepatitis C associated glomerulonephritis is an immune complex disease that occurs in 21% of patients who have HCV infection. It most commonly presents as membranoproliferative and mixed cryoglobulinemia It characterized by an indolent course in one third of patients , remission in another third and relapsing course in the remaining patients with potential progression to advanced chronic kidney disease.

mechanism of injury : Chronic Hepatitis C is primarily associated with type II cryoglobulinemia , in which the primary mechanism of injury is vasculitis that occurs via immune complex deposition.

hepatitis C virus related glomerular disease :

Type I membranoproliferative was the most common finding associated with mixed cryoglobulinemia but other forms of glomerulonephritis were associated with Hepatitis c like mesangial glomerulonephritis,focal and segmental glomerulonephritis,minimal change nephropathy,membranous nephropathy , Fibrillary glomerulonephritis,immunotactoid glomerulopathy,IgA nephropathy, vasculitic renal involvement ,poly arteritis nodosa and interstitial nephritis .

ELIGIBILITY:
Inclusion Criteria:

* it will be conducted on chronic hepatitis C patients with chronic kidney disease .
* The participants will be classified according to their estimated GFR by modified MDRD equation and
* they will be recruited from the renal unit of internal medicine, Assiut University Hospitals and assiut hepatitis viruses unit-ministry of health, Egypt.

Exclusion Criteria:

Patients will be excluded if the underlying causes of CRF are as follows:

chronic pyelonephritis,obstructive uropathy,Polycystic kidney disease,Patients with ESRD on regular hemodialysis,patients with advanced liver cirrhosis,hepatocellular carcinoma,Patients on steroids or immunosuppressive drugs and Solitary kidney.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: prospective observational study
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2018-11 (Estimated); Primary Completion 2019-10 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
prevalence of histopathological pattern in patients with hepatitis C virus | one year
  prevalence of histopathological pattern in patients with hepatitis C virus

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Tohammy, PhD, Study Director — Faculty of medicine , internal medicine ,Assuit university
Locations (1):
- Assuit University, Asyut, Egypt